CLINICAL TRIAL: NCT01390129
Title: Remote Ischemic Preconditioning in Aortic Valve Surgery (RIP-Valve)
Brief Title: Remote Ischemic Preconditioning in Aortic Valve Surgery
Acronym: RIP-Valve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOI 2010-07
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Experimental)
  Interventions: Procedure: Control
- Remote ischemic preconditioning (Active Comparator)
  Interventions: Procedure: Remote ischemic preconditioning

INTERVENTIONS:
Procedure: Control — Deflated blood pressure cuff placed on upper arm for 30min
  Arms: Control
Procedure: Remote ischemic preconditioning — Blood pressure cuff placed on upper arm and inflated to 200 mmHg for 5 min and then deflated for 5 min. This cycle is initiated before aortic clamping and repeated 3 times in total
  Arms: Remote ischemic preconditioning

SUMMARY:
RIP-VALVE is a randomized, single blinded study that will test the hypothesis that remote ischemic preconditioning initiated before surgery reduces post-operative myocardial damage in aortic valve surgery. Infarct size will be determined by 72 hours area under curve of troponin-I.

DETAILED DESCRIPTION:
The hypothesis tested in this research proposal is that remote ischemic preconditioning initiated immediately before aortic valve surgery reduces myocardial damage related to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Aortic valve surgery for aortic stenosis
* Written informed consent

Exclusion Criteria:

* Aortic valve surgery combined with CABG or an other valve surgery
* Previous Q-wave myocardial infarction or previous coronary artery bypass graft
* Coronary artery stenosis >70%
* Ejection fraction <35%
* Surgery performed in emergency
* Nicorandil ou metformin treatment within 8 days before surgery
* Patient refusal / patient not having provided written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Infarct size | 72 hours
  Infarct size as assessed by 72 hours area under curve serum troponin-I

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Prunier, MD, PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- University Hospital, Angers, Angers, France

REFERENCES:
- [Derived] Chao de la Barca JM, Bakhta O, Kalakech H, Simard G, Tamareille S, Catros V, Callebert J, Gadras C, Tessier L, Reynier P, Prunier F, Mirebeau-Prunier D. Metabolic Signature of Remote Ischemic Preconditioning Involving a Cocktail of Amino Acids and Biogenic Amines. J Am Heart Assoc. 2016 Sep 24;5(9):e003891. doi: 10.1161/JAHA.116.003891. PMID 27664804